CLINICAL TRIAL: NCT04435652
Title: A Study of QL1604 Plus Nab-paclitaxel Versus Paclitaxel for Participants With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma That Progressed After Therapy With Platinum and Fluoropyrimidine
Brief Title: A Study of QL1604 Plus Nab-paclitaxel Versus Paclitaxel in Subjects With Advanced Gastric Cancer.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1604-302
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Intervention Model Description: The first stage is a single-arm clinical trial, and the second stage is a controlled clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Cohort A (Experimental): Participants receive QL1604 and nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle. If not disease progression after 4 cycles, participants receive QL1604 monotherapy until disease progression、unacceptable toxicity or up to 2 years.
  Interventions: Drug: QL1604; Drug: Nab-paclitaxel
- Experimental: Cohort B-arm1 (Experimental): Participants receive QL1604 and nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle. If not disease progression after 4 cycles, participants receive QL1604 monotherapy until disease progression、unacceptable toxicity or up to 2 years.
  Interventions: Drug: QL1604; Drug: Nab-paclitaxel
- Experimental: Cohort B-arm2 (Experimental): Participants receive paclitaxel on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: QL1604 — 3mg/kg, D1,8,15,Q4w, IV infusion
  Arms: Experimental: Cohort A; Experimental: Cohort B-arm1
Drug: Nab-paclitaxel — 100mg/m2, D1,8,15,Q4w, IV infusion
  Arms: Experimental: Cohort A; Experimental: Cohort B-arm1
Drug: Paclitaxel — 80mg/m2, D1,8,15,Q4w, IV infusion
  Arms: Experimental: Cohort B-arm2

SUMMARY:
This is a study for participants with advanced gastric or gastroesophageal junction adenocarcinoma who had tumor progression after first-line treatment with platinum and fluoropyrimidine doublet therapy. The study will be conducted in 2 parts.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; Completely understand and know this study as well as sign the informed consent form (ICF);
2. Age ≥ 18 years and ≤ 80 years when ICF is signed;
3. Have histologically or cytologically confirmed diagnosis of locally advanced, unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma(G/GEJC).
4. Eastern Cooperative Oncology Group performance status of 0 or 1;
5. Life expectancy of at least 12 weeks;
6. Have measurable disease as defined by RECIST 1.1 as determined by the investigator;
7. Be willing to provide newly-obtained or paraffin-embedded tissue for PD-L1 and other biomarker analysis;
8. HER-2/neu negative；
9. Female subjects of childbearing potential should have a negative serum human chorionic gonadotropin(HCG) test within 7 days prior to receiving the first dose of study medication and are not breastfeeding;
10. Male and female subjects able to have children must agree to use highly effective method of contraception throughout the study and for at least 180 days after last dose.

Exclusion Criteria:

1. Has non-G/GEJC such as squamous cell carcinoma, adenosquamous carcinoma, undifferentiated gastric cancer;
2. Known allergy or hypersensitivity to QL1604/nab-paclitaxel/paclitaxel or any components used in the preparation;
3. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease disease-relieving drugs, corticosteroids or immunosuppressant）;
4. Has a diagnosis of immunodeficiency or received systemic steroid therapy （>10mg daily of prednisone or equivalent drug）or any other form of immunosuppressive therapy within 14 days prior to the planned start of study therapy；
5. Subjects who have received radiotherapy, chemotherapy, monoclonal antibodies,targeted therapy, other anti-tumor treatments,or participating in other clinical studies is less than 4 weeks before the first dose of trial treatment;
6. Has a known additional malignancy that is progressing or requires active treatment in past 3 years;
7. Subjects with known central nervous system (CNS) metastasis;
8. Has a history of pneumonitis that required steroids in past 3 years;
9. Has an active infection requiring systemic therapy；
10. Subjects with the history of Human Immunodeficiency Virus (HIV)、acquired, congenital immunodeficiency diseases、organ transplant;
11. Has hepatitis B surface antigen (HBsAg) positive and/or hepatitis B core antibody (HBcAb) positive and HBV deoxyribonucleic acid (HBV DNA) >1000 copies/mL, or hepatitis C virus antibody positive;
12. Has received a live vaccine within 30 days of the planned start of study therapy；
13. Has received prior immune checkpoint inhibitors;
14. Known psychiatric or substance abuse disorders that would interfere with the requirements of the study;
15. Subjects with uncontrollable cardiac diseases;
16. Has accompanying diseases that seriously endanger the subject's safety or affect the study by the investigator;
17. Has any condition that increases the risk, interferes with the study results by the investigator, or investigators/sponsor consider the subjects are not suitable for this trial;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AE) and serious adverse events (SAE) according to CTCAE V5.0 | Up to 90 days from last dose
  Safety and tolerability (stage 1)
The percentages of participants discontinuing or suspending the study drug due to an AE. | Up to 90 days from last dose
  Safety and tolerability (stage 1)
Overall survival（OS）（stage 2） | from the date of first dose until the date of death from any cause,assessed up to 2 years
  Overall survival is defined as time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective response rate（ORR）assessed by the investigators according to RECIST 1.1（stage 1 and 2） | up to 2 years
  Objective response rate（ORR）assessed by the investigators according to RECIST 1.1.
Disease control rate（DCR）assessed by the investigators according to RECIST 1.1（stage 1 and 2） | up to 2 years
  Disease control rate（DCR）assessed by the investigators according to RECIST 1.1.
Progression-free survival（PFS）assessed by the investigators according to RECIST 1.1（stage 1 and 2） | up to 2 years
  Progression-free survival（PFS）assessed by the investigators according to RECIST 1.1.
Tumor response rate（TRR）assessed by the investigators according to RECIST 1.1（stage 1 and 2） | up to 2 years
  Tumor response rate（TRR）assessed by the investigators according to RECIST 1.1.
Overall survival(stage 1) | from the date of first dose until the date of death from any cause,assessed up to 2 years
  Overall survival is defined as time from randomization to death due to any cause.
Area under the concentration-time curve (AUC ) following single dose administration of PD-1（stage 1 ） | through study completion, an average of 2 years
  Area under the concentration-time curve (AUC ) following single dose administration of PD-1
Peak plasma concentration (Cmax) following single dose administration of PD-1（stage 1 ） | through study completion, an average of 2 years
  Peak plasma concentration (Cmax) following single dose administration of PD-1
Steady-state trough serum concentration of multiple Dose Administration of PD-1（stage 2） | through study completion, an average of 2 years
  Steady-state trough serum concentrationof multiple Dose Administration of PD-1
Steady-state peak serum concentration of multiple Dose Administration of PD-1（stage 2） | through study completion, an average of 2 years
  Steady-state peak serum concentration of multiple Dose Administration of PD-1
Immunogenicity（stage 1 and 2） | through study completion, an average of 2 years
  The titer of anti-drug antibodies (ADA)and neutralizing antibodies(Nab).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China